CLINICAL TRIAL: NCT03925090
Title: Randomized, Placebo-controlled, Double-blind Phase II Clinical Trial of Neoadjuvant and Adjuvant Anti-PD-1 Antibody Toripalimab Immunotherapy Combined With Concurrent Chemoradiotherapy for High-risk Nasopharyngeal Carcinoma
Brief Title: Phase II Trial of Neoadjuvant and Adjuvant Anti-PD-1 Antibody Toripalimab Combined With CCRT in NPC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2019-014-01
Record Dates: First submitted 2019-03-28; First posted 2019-04-23 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant and Adjuvant Toripalimab+CCRT (Experimental): Drug: Cisplatin cisplatin 100mg/m2(every three weeks),D1,D22,D43 of intensity modulated radiotherapy Other Names: DDP Drug: Toripalimab Toripalimab 240mg every 2 weeks with a total of 2 cycles as neoadjuvant anti-PD-1 immunotherapy; Toripalimab240mg every 3 weeks with a total of 8 cycles as adjuvant anti-PD-1 immunotherapy 2 weeks after CCRT Other Names:anti-PD-1 antibody, JS001
  Interventions: Drug: Cisplatin+Toripalimab
- Neoadjuvant and Adjuvant Placebo+CCRT (Placebo Comparator): Drug: Cisplatin cisplatin 100mg/m2(every three weeks),D1,D22,D43 of intensity modulated radiotherapy Other Names: DDP Drug: placebo placebo 240mg every 2 weeks with a total of 2 cycles as neoadjuvant treatment; placebo 240mg every 3 weeks with a total of 8 cycles as adjuvant treatment 2 weeks after CCRT.
  Interventions: Drug: Cisplatin+placebo

INTERVENTIONS:
Drug: Cisplatin+Toripalimab — chemotherapy and monoclonal antibody
  Other Names: DDP+ JS001
  Arms: Neoadjuvant and Adjuvant Toripalimab+CCRT
Drug: Cisplatin+placebo — chemotherapy
  Other Names: DDP
  Arms: Neoadjuvant and Adjuvant Placebo+CCRT

SUMMARY:
This is a randomized Phase II trial to study the effectiveness and toxicity of neoadjuvant and adjuvant PD-1 antibody Toripalimab combined with concurrent cisplatin chemoradiotherapy versus cisplatin concurrent chemoradiotherapy plus placebo in treating patients with high risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China and Southeast Asia. For locoregionally advanced NPC, especially for the high risk NPC (plasma EBV DNA ≥ 1500 copies/ml), the incidence of treatment failure is still high. Although concurrent chemoradiotherapy (CCRT) can improve the treatment outcomes of these patients, approximately 25% of locoregionally advanced NPCs still develop relapse and metastasis.

Hence, there is an urgent need for novel therapies to improve survival and reduce treatment-related toxicity in NPC patients. Accumulating evidence shows that PD-1 antibody is effective for treating recurrent/metastastic NPC patients. This is a Phase II randomized trial to study the effectiveness and toxicity of neoadjuvant and adjuvant PD-1 antibody Toripalimab combined with CCRT versus CCRT plus placebo in treating patients with high risk NPC (Stage III-IVa, AJCC 8th and EBV DNA ≥ 1500 copies/ml).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III Original clinical staged as III-IVa （according to the 8th AJCC edition）
2. No evidence of distant metastasis (M0)
3. Plasm EB Virus DNA≥1500copies/ml
4. Male and no pregnant female
5. Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1
6. WBC ≥ 4×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
7. With normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN)
8. With normal renal function test ( creatinine clearance ≥60 ml/min)

Exclusion Criteria:

1. Patients have evidence of relapse or distant metastasis
2. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
3. Receiving radiotherapy or chemotherapy previously
4. The presence of uncontrolled life-threatening illness
5. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
6. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
7. Patients who have been treated with inhibitors of immune regulation (CTLA-4, PD-1, PD-L1, etc.).
8. Patients with immunodeficiency disease and history of organ transplantation.
9. Patients who have used large doses of glucocorticoids, anti-cancer monoclonal antibodies, and other immunosuppressive agents within 4 weeks.
10. HIV positive.
11. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
12. Severe, uncontrolled medical conditions and infections.
13. At the same time using other test drugs or in other clinical trials.
14. Refusal or inability to sign informed consent to participate in the trial.
15. Other treatment contraindications.
16. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.
17. Hepatitis B surface antigen (HBsAg) positive and HBVDNA ≥1000cps/ml.
18. Patients with positive HCV antibody test results can only be included in the study when the polymerase chain reaction of HCV RNA is negative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-08 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Defined as the time from randomisation to death.
Locoregional Relapse-Free Survival (LRRFS) | 2 years or until the date of the last follow-up visit.
  Defined as the time from the randomisation to documented locoregional recurrence or death due to any cause.
Distant Metastasis-Free Survival (DMFS) | 2 years
  Defined as the time from randomisation to documented distant metastasis or death due to any cause.
Objective Response Rate （ORR） | After the completion of the neoadjuvant PD-1 antibody and chemoradiotherapy treatment
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Incidence rate of adverse events (AEs) | 2 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Correlation between the plasma EBV DNA level and PFS | 2 years
  The plasma EBV DNA level of the patients will be assessed.
Correlation between pre-treatment PD-L1 expression level and PFS | 2 years
  Pre-treatment PD-L1 expression level is evaluated centrally by means of immunohistochemical testing.
Correlation between the percentage of tumor-infiltrating lymphocytes (TILs) and PFS | 2 years
  TILs are lymphoid cells (T cells) that infiltrate solid tumors (intra-tumoral TILs) and stroma (stromal TILs), which play important roles in the tumor microenvironment.
Change of QoL (quality of life) | 1 year
  QoL scores were assessed by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before neoadjuvant PD-1 antibody, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy.
Number of subjects with major pathologic response (MPR) | 21-28 days
  Major pathologic response rate (MPR) is defined as > 90% decrease in viable tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Overall Study Officials Mai, MD,PhD, Principal Investigator — Sun Yat-Sen University Cancer Cente
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Background] Langendijk JA, Leemans CR, Buter J, Berkhof J, Slotman BJ. The additional value of chemotherapy to radiotherapy in locally advanced nasopharyngeal carcinoma: a meta-analysis of the published literature. J Clin Oncol. 2004 Nov 15;22(22):4604-12. doi: 10.1200/JCO.2004.10.074. PMID 15542811
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Twu CW, Wang WY, Chen CC, Liang KL, Jiang RS, Wu CT, Shih YT, Lin PJ, Liu YC, Lin JC. Metronomic adjuvant chemotherapy improves treatment outcome in nasopharyngeal carcinoma patients with postradiation persistently detectable plasma Epstein-Barr virus deoxyribonucleic acid. Int J Radiat Oncol Biol Phys. 2014 May 1;89(1):21-9. doi: 10.1016/j.ijrobp.2014.01.052. PMID 24725686
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Leung SF, Zee B, Ma BB, Hui EP, Mo F, Lai M, Chan KC, Chan LY, Kwan WH, Lo YM, Chan AT. Plasma Epstein-Barr viral deoxyribonucleic acid quantitation complements tumor-node-metastasis staging prognostication in nasopharyngeal carcinoma. J Clin Oncol. 2006 Dec 1;24(34):5414-8. doi: 10.1200/JCO.2006.07.7982. PMID 17135642
- [Background] Lin JC, Wang WY, Chen KY, Wei YH, Liang WM, Jan JS, Jiang RS. Quantification of plasma Epstein-Barr virus DNA in patients with advanced nasopharyngeal carcinoma. N Engl J Med. 2004 Jun 10;350(24):2461-70. doi: 10.1056/NEJMoa032260. PMID 15190138
- [Background] Economopoulou P, Agelaki S, Perisanidis C, Giotakis EI, Psyrri A. The promise of immunotherapy in head and neck squamous cell carcinoma. Ann Oncol. 2016 Sep;27(9):1675-85. doi: 10.1093/annonc/mdw226. Epub 2016 Jul 5. PMID 27380958
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Weber JS, Kudchadkar RR, Yu B, Gallenstein D, Horak CE, Inzunza HD, Zhao X, Martinez AJ, Wang W, Gibney G, Kroeger J, Eysmans C, Sarnaik AA, Chen YA. Safety, efficacy, and biomarkers of nivolumab with vaccine in ipilimumab-refractory or -naive melanoma. J Clin Oncol. 2013 Dec 1;31(34):4311-8. doi: 10.1200/JCO.2013.51.4802. Epub 2013 Oct 21. PMID 24145345
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Okazaki T, Chikuma S, Iwai Y, Fagarasan S, Honjo T. A rheostat for immune responses: the unique properties of PD-1 and their advantages for clinical application. Nat Immunol. 2013 Dec;14(12):1212-8. doi: 10.1038/ni.2762. PMID 24240160
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Schoenfeld JD. Immunity in head and neck cancer. Cancer Immunol Res. 2015 Jan;3(1):12-7. doi: 10.1158/2326-6066.CIR-14-0205. PMID 25568068
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Hsu MC, Hsiao JR, Chang KC, Wu YH, Su IJ, Jin YT, Chang Y. Increase of programmed death-1-expressing intratumoral CD8 T cells predicts a poor prognosis for nasopharyngeal carcinoma. Mod Pathol. 2010 Oct;23(10):1393-403. doi: 10.1038/modpathol.2010.130. Epub 2010 Jul 23. PMID 20657553
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Labrijn AF, Buijsse AO, van den Bremer ET, Verwilligen AY, Bleeker WK, Thorpe SJ, Killestein J, Polman CH, Aalberse RC, Schuurman J, van de Winkel JG, Parren PW. Therapeutic IgG4 antibodies engage in Fab-arm exchange with endogenous human IgG4 in vivo. Nat Biotechnol. 2009 Aug;27(8):767-71. doi: 10.1038/nbt.1553. Epub 2009 Jul 20. PMID 19620983
- [Background] Liu J, Blake SJ, Yong MC, Harjunpaa H, Ngiow SF, Takeda K, Young A, O'Donnell JS, Allen S, Smyth MJ, Teng MW. Improved Efficacy of Neoadjuvant Compared to Adjuvant Immunotherapy to Eradicate Metastatic Disease. Cancer Discov. 2016 Dec;6(12):1382-1399. doi: 10.1158/2159-8290.CD-16-0577. Epub 2016 Sep 23. PMID 27663893
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Derived] Liu SL, Li XY, Yang JH, Wen DX, Guo SS, Liu LT, Li YF, Luo MJ, Xie SY, Liang YJ, Sun XS, Yang ZC, Lv XF, Luo DH, Li JB, Liu Q, Wang P, Guo L, Mo HY, Sun R, Yang Q, Lan KQ, Jia GD, Li R, Zhao C, Xu RH, Chen QY, Tang LQ, Mai HQ. Neoadjuvant and adjuvant toripalimab for locoregionally advanced nasopharyngeal carcinoma: a randomised, single-centre, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2024 Dec;25(12):1563-1575. doi: 10.1016/S1470-2045(24)00504-7. Epub 2024 Nov 7. PMID 39522541